CLINICAL TRIAL: NCT06843070
Title: Comparison of the Effects of Sacral Erector Spinae Plane Block and Dorsal Penile Block on Postoperative Pain in Circumcision Operations
Brief Title: Comparison of the Effects of Sacral Erector Spinae Plane Block and Dorsal Penile Block on Postoperative Pain in Circumcision Procedures
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Konya City Hospital (Other)
Responsible Party: Principal Investigator, Yasin Tire, MD, Anesthesiology and Reanimation, Konya City Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Study Pedsac
Record Dates: First submitted 2025-02-09; First posted 2025-02-24 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Postoperative Analgesia
Keywords: Pediatric Regional Anesthesia; Sacral Erector Spinae Plane Block; Postoperative Analgesia in Circumcision

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The single-blind design of this study keeps some participants unaware of their group designations to reduce bias.
  Evaluators: Clinicians collecting postoperative data and assessing pain will be blinded to patient group allocation. This eliminates subjective FLACC pain scoring and postoperative analgesia evaluation. A blinded observer will measure FLACC pain at 0, 1, 2, 4, and 6 hours postoperatively.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group P (Penile Block) (Active Comparator): Patients who underwent Dorsal Penile Block after circumcision surgery
  Interventions: Procedure: PENILE BLOCK ARM
- Group S (Sacral ESP Block) (Active Comparator): Patients who underwent Sacral Erector Spinae Plane Block after circumcision surgery
  Interventions: Procedure: SACRAL ESP BLOCK ARM

INTERVENTIONS:
Procedure: PENILE BLOCK ARM — P arm: Patients who underwent Dorsal Penile Block after circumcision surgery
  Arms: Group P (Penile Block)
Procedure: SACRAL ESP BLOCK ARM — S arm: Patients who underwent Sacral Erector Spinae Plane Block after circumcision surgery
  Arms: Group S (Sacral ESP Block)

SUMMARY:
Egypt performed circumcision in 2300 BC, although its origin is unknown. Some societies use circumcision for health, whereas others do it for religious and cultural reasons . Our competent pediatric surgeons perform circumcisions without ultrasonography using midazolam (0.1 mg/kg) premedication and penile block. In addition to penile block, general anesthesia is given using sevoflurane, ketamine, fentanyl, and propofol, depending on age and weight, for intraoperative anesthesia and analgesia. Penis procedures are frequently simple (phimosis, circumcision), but the pain is significant and long-lasting, affecting young patients' postoperative recovery. The topic of analgesia remains relevant and important in anesthesia practice. Early patient mobilization and discharge are crucial. Pediatric opioid use is questioned due to adverse effects include somnolence, vomiting, and respiratory depression. The advent of ultrasound-guided nerve blocks has revolutionized regional anesthesia in pediatrics. Many upper and lower abdominal operations use truncal blocks with good success and patient safety. Since its applicability, ease of anatomical approach, distance to the medulla spinalis and surgical site, and minimal risk of infection, sacral ESP block has become a popular method for youngsters. Postoperative pain trials demonstrate it works well.

DETAILED DESCRIPTION:
Although it is not known exactly where it was first performed, there is evidence that the Egyptians performed circumcision in 2300 BC. While circumcision is performed for health reasons in some societies, it is a traditional, religious and cultural practice in some. In our clinic, circumcision cases are performed with anesthesia monitoring and premedication with midazolam (0.1 mg/kg) followed by penile block, which is our clinical practice, by experienced pediatric surgeons who perform the surgical procedure without the use of ultrasound. In addition to penile block in standard practice, general anesthesia is applied to patients with sevoflurane, ketamine, fentanyl and propofol, depending on the patient's age and weight, depending on the need for intraoperative anesthesia and analgesia. Postoperative pain after surgeries on the penis is a problem that directly affects postoperative recovery in young patients because the surgical procedure itself is often minor (treatment of phimosis, circumcision), whereas the pain produced is both severe and long-lasting.

The need for analgesia is a topic that always occupies anesthesia practice and maintains its relevance. It is vital to ensure early mobilization and discharge of patients. Many side effects, including somnolence, vomiting and respiratory depression, call into question the use of opioids in pediatrics.

Today, the use of ultrasound-guided nerve block has resulted in a revolutionary change in the field of regional anesthesia in pediatrics. Many truncal blocks are used with a high success rate in both upper and lower abdominal surgeries and have become standard in terms of patient safety.

Sacral ESP block, especially applied in children, has become an increasingly important technique due to its advantages such as applicability, ease of anatomical approach, distance to the medulla spinalis and surgical site, and low risk of infection. In addition, studies have shown that it is quite effective in postoperative pain.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria of the patients: Age between 7-12 years, ASA Physical Status 1 and 2, circumcision surgery, general anesthesia, planned hospital stay of at least 24 hours.

Exclusion Criteria:

* Exclusion criteria were defined as patients whose family or personal consent could not be obtained for the study, Asa 3 and above cases, patients in the study age group who will undergo emergency surgery, patients with serious hematopoietic system, cardiovascular, liver or kidney disease, patients receiving anticoagulation therapy, patients with sensitivity to regional anesthetic agents and patients who have previously undergone penile surgery.

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2025-02-25 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2025-12-25 (Estimated)

PRIMARY OUTCOMES:
PRIMARY OUTCOME | Postoperative ''0 hour, 1. hour, 2.hour, 4.hour, 6 hour
  The primary outcome variable of the study will be the FLACC pain score transferred to the pacu after surgery. Patients will be assessed for pain with the FLACC pain scale at 30-minute intervals throughout the pacu stay and at 0, 1, 2, 4 and 6 hours until discharge from the hospital.

SECONDARY OUTCOMES:
SECONDARY OUTCOME | postoperative '' before the discharge''
  As a secondary outcome variable, a simple pain scale was explained to parents to fill in the rating sheet as a measure of satisfaction with postoperative pain (0 = no pain/child calm; 1 = minimal pain/child irritable; 2 = mild pain/child consolable; and 3 = severe pain/child inconsolable).

CONTACTS AND LOCATIONS:
Locations (1):
- Yasin Tire, Konya, Meram, Turkey (Türkiye)